CLINICAL TRIAL: NCT02672059
Title: Pain In Neuropathy Study
Acronym: PINS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: University of Oxford (Other); Imperial College London (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 10/H0706/035; 9755 (Other: UK Clinical Research Network)
Record Dates: First submitted 2016-01-05; First posted 2016-02-03 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Neuropathy; Neuropathic Pain; Chronic Pain; Carpal Tunnel Syndrome; Peripheral Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia; Chronic Pain; Carpal Tunnel Syndrome; Peripheral Nervous System Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1. We will collect blood samples (30mls) from each subject, which will be stored at -800C in a locked freezer. All samples will eventually be transported to King's College for storage in compliance with The Human Tissues Act. DNA will be taken for studies in genetics polymorphisms or mutations within genes which may modify the risk of a person developing a neuropathic pain and/or the severity of neuropathic pain, if and only if patients agree. Genetic analysis will be strictly restricted to the neuropathic pain field, and data will be anonymised after blood has been taken from patients. If blood chemistry and HbA1c is not available from primary care, these will also be checked. We will also assess new potential metabolic biomarkers in the serum of patients that can shed a light into mechanisms for the development of neuropathy and pain.
  2. IENFD assessed via one 3mm skin punch biopsies performed 10 cm above lateral malleolus.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peripheral Neuropathy: Patients with peripheral neuropathy (observational study, no interventions)
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No intervention

SUMMARY:
In the context of peripheral neuropathy, we will aim to elucidate correlates between sensory symptoms and:

* Sensory nerve dysfunction.
* Cutaneous small nerve fibre innervation density.
* Psychological co-morbidity.
* Circadian rhythm disturbance co-morbidity.
* Functionality and Quality of life.
* Patterns of human brain activity in a subset of patients that consent to participate in the FMRI (functional magnetic resonance imaging) component of PINS.

  2. We will also collect blood samples in this phenotyped cohort of patients. These blood samples coupled with detailed phenotype data will investigate potential gene associations only in the development of painful neuropathy.

  3. Knowledge gained from the study will be used to aid the further development of pain questionnaires, designed to detect patients with painful neuropathy.

  4.Knowledge gained from the study will be invaluable in informing on-going investigations of painful peripheral neuropathy in animal models, both in our laboratory and others.

DETAILED DESCRIPTION:
Very little is currently known about why some patients with peripheral neuropathy develop neuropathic pain, whilst others do not. It is anticipated that this study will begin to identify features of the peripheral neuropathy, which are and are not, associated with the development and intensity of neuropathic pain and therefore begin to elucidate factors, which underlie pain. We will also compare findings in neuropathies resulting from diverse aetiologies including diabetes, HIV and idiopathic axonal neuropathies in order to investigate, whether there are differences in pain symptomatology, NCS, QST, patterns of evoked brain activity and small fibre dysfunction in these different contexts.

We would like to answer the following question:

'In patients suffering from peripheral neuropathy what are the relationships between pain symptomatology and peripheral sensory dysfunction, intraepidermal nerve fibre density (IENFD) and psychological, and circadian rhythm co-morbidity as well as in everyday functionality?

1.2.1 Quantitative sensory testing (QST) and neuropathic pain.

Nerve conduction studies (NCS) predominantly assess large fibre function and indeed in the context of small fibre neuropathy are often normal. We propose to assess the utility of two relatively non-invasive tools, which are routinely used, both in our practice and elsewhere, to assess small fibre dysfunction: quantitative sensory testing (QST) and intraepidermal nerve fibre density (IENFD). There have been studies examining both of these in the context of neuropathy, but the exact relationship of these measures to abnormalities to pain, quality of life and psychological state is largely unknown.

QST is a method for accurately determining sensory thresholds in human skin and is particularly useful for determining dysfunction in the nociceptive smaller diameter nerve fibres, although the precise utility of QST in routine clinical neuropathic pain management perhaps requires some further evaluation. There is also increasing interest in using QST in combination with assessment of pain descriptors to give insights into the underlying pathophysiological mechanisms of chronic pain. For example, the presence of brush evoked dynamic allodynia indicates sensitisation at the spinal level. Although QST is widely used as an assessment tool for small fibre function and sensory phenotype in neuropathies associated with pain often only certain individual components have been measured (e.g. thermal and vibration thresholds as opposed to the full battery of tests required to give the complete sensory assessment). Previous studies have also suggested that patients with painful neuropathy may also display hyperalgesia to mechanical and thermal suprathreshold stimuli, however these studies have contained relatively small numbers of subjects. We will therefore further characterise this phenomenon by conducting additional suprathreshold mechanical and thermal stimuli according to a method previously described, in addition to the standard German Neuropathic Pain Network QST protocol, and also we will include variations in ambient temperature (in the range of 10 to 35 °C) to assess if characteristics related to the sensory testing eventually change.

1.2.2 Intra-epidermal nerve fibre density (IENFD) and neuropathic pain.

Measurement of IENFD is a relatively simple assay which can be performed in relatively innocuous 3mm punch biopsies of skin, a routine dermatological investigation. Its utility in the assessment of small fibre function in peripheral neuropathies is clear. Peripheral neuropathies of diverse aetiologies are associated with reduced epidermal innervation density however the exact relationship of this reduction to pain and pain co-morbidities requires proper evaluation. Residual skin tissue will be stored in compliance with The Human Tissue Act, for further biochemical analysis.

1.2.3 Nerve Conduction Studies Axon Reflex and Neuropathic Pain Characteristically, different types of peripheral neuropathy exhibit patterns of demyelination or axonopathy in large fibres. The rationale for the procedure in this study is to discard other pathologies that may account as the main etiology causing pain in the context of a peripheral neuropathy. Guillain-Barre Syndrome, Chronic Inflammatory Demyelinating Polyradiculoneuropathy, Vasculitic Neuropathies and others can account for both neuropathy and pain allowing us to make the sample more homogeneous. Nerve conduction studies are usually safe procedures in which the indemnity of the axon and its myelin sheath are tested using external electrical stimuli. As a part of the protocol we have these tests . As a part of the study, Electromyography (EMG) will not be included either.

If NCS have been performed as part of the patients routine medical care these results will be recorded.

As a further means of assessing the physiological integrity of C fibers in patients suffering from carpal tunnel syndrome we will elicit an axon reflex. This reflex involves the transcutaneous application of agents such as histamine via iontophoresis (electrical current). The histamine will stimulate the peripheral nerve endings of the small diameter C fibres. Their stimulation induces a vasodilatation, which is visible as a flare response of the skin. The evaluation of the extent of the flare response is used as an indication of the integrity of the small diameter C fibre population.

1.2.4 Psychological co-morbidity, quality of life and neuropathic pain

Whilst some studies have examined aspects of pain in the context of peripheral neuropathy, these do not go beyond more than simple measurement of pain intensity or sensory characteristics and there is only a limited literature which has explored the interactions between pain, psychological status and quality of life. Neuropathic pain in general is associated with multiple psychological problems which impact upon quality of life. These include circadian rhythm disturbances (e.g. sleeping difficulty: moderate to severe in 60% of patients), lack of energy (55%), drowsiness (39%) and difficulty in concentration (36%); similar findings have been specifically documented in diabetic neuropathy. Severe to moderate depression and anxiety also occur in about 30% of neuropathic pain patients. In general, beliefs and fears concerning the pain and its implications contribute substantially to determining mood and behaviour. Since neuropathic pain is relatively common in the context of peripheral neuropathy the question arises as to what extent pain is the driver of these co-morbidities - the answer to this is not known, but large randomised controlled trials of analgesic interventions in neuropathic pain states indicate that as pain intensity reduces so does the severity of these co-morbidities. To answer this question we will first need to identify specific tools for the measurement of neuropathic pain co-morbidity in the context of peripheral neuropathy this is one of the aims of this proposal and we will evaluate a variety of existing assessment tools. Another issue is that it is likely that psychological co-morbidity influences the self reporting of pain intensity, which is a usual primary outcome measure in clinical trials of neuropathic pain analgesic agents.

We will use a battery of psychological instruments to determine the psychological and quality of life in those subjects with peripheral neuropathy and identify differences between those who do and do not suffer from neuropathic pain.

We will also attempt to further validate a number of neuropathy screening and assessment tools; the Brief Peripheral Neuropathy Screen (BPNS) and the Utah Early Neuropathy Scale (UENS). The BPNS and UENS tools has been previously evaluated in the context of HIV and diabetic neuropathy respectively, however our study would provide additional invaluable information in the light of both QST and IENFD findings in the context of axonal polyneuropathy resulting from diverse aetiologies.

1.2.4 Blood samples

We will collect blood samples (30mls) from each subject, which will be stored at -80C in a locked freezer. This coupled with the detailed phenotype data collected, will inform studies investigating potential genetic associations in the development of neuropathic pain. A serum sample will also be stored for the consideration of future biomarker studies.

1.2.5 Imaging human brain activity in a subset of PINS participants

The advent of functional imaging techniques allowed researchers to begin to look within the human brain to observe what pain looks like in the brain. Initially, pain imaging research determined that pain is not processed by a single brain region but instead engages several distributed cortical areas. The group of brain regions that are most active during pain are commonly referred to as the 'pain matrix'. This includes: primary and secondary somatosensory cortices (SI, SII), insular, anterior cingulate, and prefrontal cortices and the thalamus. However, pain is not purely a sensory event but is also reflective of how the person feels about their pain. Factors that vary widely across a population such as memories, emotion, pathology, genetics, and cognitive factors all directly affect how an individual experiences pain. Because of this, the pain matrix provides an incomplete picture of what is happening in the brain during pain. Pain imaging studies have begun to validate this perspective. For example, Derbyshire et al. showed activation of the key pain matrix regions even when subjects were not in pain. From a study looking at chronic pain sufferers, Baliki et al. showed that a series of other key brain regions were active that were outside the pain matrix. It is essential for brain imaging research to update the notion of the 'pain matrix' to account for these inconsistencies. Therefore, in this study we would like to see which areas of the brain are activated when the peripheral markers of the polyneuropathy are targeted by a range of noxious and non-noxious stimulations, so that we can determine the key brain regions involved in pain processing.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are ≥18 years of age who have a diagnosis of peripheral neuropathy based on a prior clinical assessment combined with supportive clinical investigations such as abnormal nerve conduction studies, reduced intraepidermal nerve or abnormal findings on quantitative sensory testing.
* If supportive clinical investigations (as described above) are not available at entry into the study a neuropathy disability scale ≥3 (Pham et al., 2000).
* And patients with symptoms highly suggestive of neuropathy that in the judgement of the clinical researcher are suitable for the study even if they do not fulfill other inclusion criteria.
* Patients who do not fulfill any of the exclusion criteria.

Exclusion Criteria:

* Subjects who are pregnant.
* Subjects with insufficient command of English to obtain consent from or to complete the study questionnaires.
* Subjects with insufficient mental capacity to obtain consent from or complete study questionnaires.
* Subjects with concurrent severe psychological or psychiatric disorders.
* Patients with moderate to severe pain form other causes that may confound assessment or reporting of pain (eg. spinal canal stenosis).
* Patients with central nervous lesions, which may complicate somatosensory testing.
* Who is in the opinion of the investigator unsuitable for participation in the study.
* Skin biopsies will not be conducted on patients that are anticoagulated or who have any other contra-indication to skin biopsy (if patients decline a skin biopsy they will NOT be excluded from the study).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with peripheral neuropathies associated with diabetes, carpal tunnel syndrome or others.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2011-02; Primary Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of neuropathy | Day 1
  Toronto Clinical Scoring System of 4

SECONDARY OUTCOMES:
Demographics | Day 1
  Main demographic visits
Detailed medical history | Day 1
  Past clinical records of patients relevant to the current disease status
7-days pain diary | Day 1
  Patients will have 7-days pain diaries with a numeric rating scale from 0 to 10
Pain related anxiety | Day 1
  Patients will answer the Pain Anxiety Symptoms Scale (PASS-20)
Measures of quality of life | Day 1
  Patients will answer the 36-Item Short Form Survey -quality of life questionnaire-
Measures of sleep interference | Day 1
  Sleep quality is assessed through the use of questionnaires
Nerve Conduction Studies | Day 1
  Neurophysiology will be conducted to assess nerve integrity
Sensory Thermal Thresholds | Day 1
  Thermal thresholds will be measured in degrees centigrade
Sensory Mechanical Detection Thresholds | Day 1
  Mechanical Detection Thresholds will be measured in millinewtons
Intra-Epidermal Nerve Fibre density | Day 1
  Measurement of nerve fibres in the skin of patients - leg or finger-
Blood samples - DNA | Within 6 months of visit
  Blood samples coupled with detailed phenotype data will investigate potential gene associations in the development of painful neuropathy
Blood samples - RNA | Within 18 months of visit
  Blood samples coupled with detailed phenotype data will investigate potential blood markers associations in the development of painful neuropathy
Blood samples - Serum | Within 18 months of visit
  Blood samples coupled with detailed phenotype data will investigate potential blood markers associations only in the development of painful neuropathy
Synovium tissue collection for RNA | Within 18 months of visit
  Synovium from around the nerve and tendons coupled with detailed phenotype data will investigate potential blood markers associations only in the development of painful neuropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Nuffield Department of Clinical Neurosciences, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Phillips TJC, Brown M, Ramirez JD, Perkins J, Woldeamanuel YW, Williams ACC, Orengo C, Bennett DLH, Bodi I, Cox S, Maier C, Krumova EK, Rice ASC. Sensory, psychological, and metabolic dysfunction in HIV-associated peripheral neuropathy: A cross-sectional deep profiling study. Pain. 2014 Sep;155(9):1846-1860. doi: 10.1016/j.pain.2014.06.014. Epub 2014 Jun 26. PMID 24973717
- [Result] Schmid AB, Bland JD, Bhat MA, Bennett DL. The relationship of nerve fibre pathology to sensory function in entrapment neuropathy. Brain. 2014 Dec;137(Pt 12):3186-99. doi: 10.1093/brain/awu288. Epub 2014 Oct 27. PMID 25348629
- [Result] Ramirez JD, Barnes PRJ, Mills KR, Bennett DLH. Intermediate Charcot-Marie-Tooth disease due to a novel Trp101Stop myelin protein zero mutation associated with debilitating neuropathic pain. Pain. 2012 Aug;153(8):1763-1768. doi: 10.1016/j.pain.2012.05.015. Epub 2012 Jun 16. PMID 22704856
- [Result] Segerdahl AR, Xie J, Paterson K, Ramirez JD, Tracey I, Bennett DLH. Imaging the neural correlates of neuropathic pain and pleasurable relief associated with inherited erythromelalgia in a single subject with quantitative arterial spin labelling. Pain. 2012 May;153(5):1122-1127. doi: 10.1016/j.pain.2011.12.012. Epub 2012 Feb 24. PMID 22365309
- See also: A team at the University of Oxford would like to recruit people aged over 18 who have diabetes and neuropathy to a study of the causes of neuropathic pain. Their findings could inform the development of new therapies. (Recruiting until June 2017) — https://www.diabetes.org.uk/Research/Take-part-in-research/